CLINICAL TRIAL: NCT01776281
Title: Effects of Kangaroo Mother Care Among LBW and Preterm Infants:A Randomized Control Trial in Karachi
Brief Title: Effects of Kangaroo Mother Care Among Low Birth Weight (LBW) and Preterm Infants
Acronym: KMC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ms Seema Hyderali, Student, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHyderali
Record Dates: First submitted 2013-01-22; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: LBW; Preterm
Keywords: effects; KMC; LBW; preterm; temperature; breastfeeding; secondary hospitals
MeSH Terms: conditions — Premature Birth; Breast Feeding | interventions — Kangaroo-Mother Care Method; Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kangaroo Mother Care (Experimental): Other than routine clinical care per hospital policy. Infants will receive skin-to-skin contact for minimum one hour daily during hospital stay and at home till one month.
  Interventions: Behavioral: Kangaroo Mother Care
- Standard Care (Active Comparator): Routine incubator or cot care with breastfeeding support from nurses as per policy.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Kangaroo Mother Care
  Arms: Kangaroo Mother Care
Behavioral: Standard Care
  Arms: Standard Care

SUMMARY:
- Hypothermia, infections ,and ineffective breastfeeding are some of the commonest causes of deaths among premature and low birth weight LBW infants. Even if the infants are born in facilities, incidences of cold stress are possible due to insufficient resources, space and incompetent practices to manage hypothermia in the immediate postnatal period. Kangaroo Mother Care is a well-known intervention to address the issues related to preterm births, such as hypothermia, infection and prolong hospitalization.Besides significant outcome of KMC interventions for preterm infants, no interventional study has been found in literature in Pakistani context. Looking at the potential benefits of KMC in reducing the related complications of prematurity, the study aims to identify the effectiveness of KMC among preterm and LBW infants born in secondary hospital of Aga khan University hospitals.

Hypothesis I Ha: KMC is effective in reducing the incidences of hypothermia among preterm and LBW infants as compared to the usual care.

Hypothesis II Ha: There is a difference in breastfeeding behavior and breastfeeding outcome among experimental and control group.

Secondary Hypothesis Hypothesis I Ha: There is an association between KMC and frequency of suspected infections during hospitalization.

Hypothesis II Ha: There is a difference in length of stay among experimental group and control group.

Hypothesis III Ha: There is a relationship between KMC and weight gain of infants till four weeks.

Hypothesis IV Ha: There is difference in rate of hypothermia among experimental group and control after discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Any preterm neonates (< 37 weeks of gestation by maternal dates)
* Low birth weight infants less than 2500 gm.

Exclusion Criteria:

* Infants with brain hemorrhage, congenital abnormalities.
* Infants needed double phototherapy.

Exclusion of Mother:

Mothers with severe depression, sickness with intensive care requirements. Mother who refused to participate. Mothers who delivered live multiple babies.

Ages: 1 Day to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Breastfeeding outcomes | 30 days
  Comparison of breastfeeding frequency per day, method of feeding. (partial/ exclusive)in hospital and at home.
  Breastfeeding behaviour by using preterm Infants breastfeeding behaviour Scale(PIBBS).
  Follow-up till one months by calling and record keeping of breastfeeding status.

SECONDARY OUTCOMES:
Rate of Infection | 1-2 weeks(During hospital stay)
  frequency of presume sepsis and need for antibiotics.
length of stay | 1-2 weeks
  Total days in hospital during the recruitment period.
weight gain | 30 days
  After discharge observation for weight gain in Follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Rozina Karmaliani, PhD, Study Director — Aga Kahn University School of Nursing and Midwifery; Zulfiqar Bhutta, Study Director — AKUH
Locations (1):
- Seema Hyderali, Karachi, Sindh, Pakistan